CLINICAL TRIAL: NCT04014491
Title: The Effects of Scapular Control and Strengthening Training on Neuromuscular Control and Corticospinal System in Overhead Athletes With Shoulder Impingement Syndrome
Brief Title: The Effects of Exercise Training on Corticospinal System in Overhead Athletes With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM108043F
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Shoulder Impingement Syndrome; Transcranial Magnetic Stimulation; Central Nervous System; Biomechanical Phenomena
Keywords: Shoulder impingement syndrome; Transcranial magnetic stimulation; Corticospinal system; Scapular control exercise; Kinematics
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scapula control exercise (Experimental): Subjects will perform three exercises with EMG biofeedback and verbal cues. Three exercises are elevation in scapular plane, sidelying external rotation and dynamic hug plus
  Interventions: Procedure: Scapula control exercise
- Scapula strengthening exercise (Experimental): The subjects in the scapular strengthening group will be asked to perform the three exercises the same as scapula control exercise group and with the same number of trials but without any EMG biofeedback and oral cues of movement or posture correction.
  Interventions: Procedure: scapular strengthening exercise
- Healthy subject group (Other): Healthy subjects will be included to compare the differences in corticospinal system between healthy subjects and subjects with shoulder impingement syndrome, so this group will not receive any treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: Scapula control exercise — To perform arm elevation in the scapular plane, subjects will be first asked to correct scapular resting posture in sitting with EMG biofeedback. Then the subjects will be instructed to do elevation in the scapular plane, side lying external rotation and dynamic hug plus with control of the scapula by EMG feedback and verbal cues
  Arms: Scapula control exercise
Procedure: scapular strengthening exercise — The subjects in the scapular strengthening group will be asked to perform these three exercises the same as scapula control group and with the same number of trials but without any EMG biofeedback and oral cues of movement or posture correction.
  Arms: Scapula strengthening exercise
Other: No intervention — No intervention
  Arms: Healthy subject group

SUMMARY:
Shoulder impingement syndrome is the most common shoulder disorder in overhead athletes. It describes a mechanical compression of subacromial bursa and rotator cuff tendons during arm movement, which results in pain and injuries. Most of previous studies focus on investigating motor performance in individuals with shoulder impingement syndrome and found altered scapular kinematics and muscle activation may contribute to the impingement. Recently few studies found changes in the central nervous system, decreases in corticospinal excitability and increases in inhibition in scapular muscles, by using transcranial magnetic stimulation (TMS). Although more studies are still needed to investigate the changes in central nervous system in the individuals with impingement syndrome, the changes in central nervous system are believed to be associated with the deficits of impingement syndrome. However, the exercise protocols for the impingement syndrome are usually designed to restore scapular kinematics and muscle activation, including scapular muscle strengthening exercise and scapular control exercise. To our knowledge, no study has investigated whether these exercise protocols can reverse these changes in the corticospinal system. The objectives of this proposal are to understand neuromuscular and neurophysiological mechanisms of the scapula-focused exercise protocols to improve the effectiveness of treatment. The study aims to investigate the effects of scapular muscle strengthening training and scapular control training on the scapular kinematics, muscle activation and corticospinal system. The study also aims to investigate whether any other cortical mechanisms are also affected by the shoulder impingement syndrome. We will recruit 70 overhead athletes with shoulder impingement syndrome and 22 healthy control athletes. Subjects with shoulder impingement syndrome will randomly receive either scapular muscle strengthening or scapular control training. When performing the exercise, subjects in the scapular control training group will receive electromyography feedback and cues but those in the strengthening training group will not. Immediate effects of these two training protocols on scapular kinematics, muscle activation, and neurophysiological measures will be tested before and after the training. Neurophysiological measures will be tested by TMS, including corticospinal excitability, cortical inhibition, intracortical inhibition, and intracortical facilitation.

ELIGIBILITY:
Inclusion Criteria: (patients of shoulder impingement)

1. Practice overhead exercise more than six hours a week,
2. Aged 20 to 40 years old,
3. Have shoulder pain localized at the anterior or lateral aspect of shoulder more than two weeks,
4. Have obvious medial border prominence of the scapula at 90° of arm elevation,
5. Have shoulder impingement syndrome, which is confirmed by having at least two of the following: (a) positive Neer test, (b) positive Hawkins sign, (c) positive empty can test, (d) positive resisted external rotation test, and (e) tenderness of the rotator cuff tendons

Inclusion Criteria: (healthy subjects)

1. Practice overhead exercise more than six hours a week,
2. Aged 20 to 40 years old,
3. Not have a history of shoulder or neck pain or injury.

Exclusion Criteria (patients of shoulder impingement and healthy subjects)

1. Have a history of dislocation, fracture, or surgery of upper extremity,
2. A history of direct contact injury to the neck or upper extremities within the past 12 months,
3. A concussion within the past 12 months or a history of three or more concussions,
4. Brain injury and neurological impairment,
5. History of frequent headache or dizziness,
6. Contraindications to the use of TMS, assessed with a safety screening questionnaire, including pregnancy, history of seizure, epilepsy and syncope, having cochlear implant, having medal implant and taking anti-depressant medication.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Neurophysiological measures - Active motor threshold | Immediately after the intervention
  Active motor threshold (AMT) will be described with the percentage (%) of maximum stimulator output (MSO).
Neurophysiological measures - Motor evoked potential | Immediately after the intervention
  Motor evoked potential (MEP) will be described with millivolt (mV).
Neurophysiological measures - Cortical silent period | Immediately after the intervention
  Cortical silent period (CSP) will be measured with millisecond (ms).
Neurophysiological measures - Short interval cortical inhibition | Immediately after the intervention
  Short interval cortical inhibition (SICI) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is below 5 ms
Neurophysiological measures - Intra-cortical facilitation | Immediately after the intervention
  Intra-cortical facilitation (ICF) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is above 5 ms

SECONDARY OUTCOMES:
Scapular kinematics | Immediately after the intervention
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapula plan elevation at 30°, 60°, 90°, and 120°, will be calculated and will be described with degree (°).
Scapular muscles activation | Immediately after the intervention
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, and serratus anterior will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- Yin-Liang Lin, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No